CLINICAL TRIAL: NCT02117479
Title: A Randomized, Double-Blind, Phase 3 Study of the JAK1/2 Inhibitor, Ruxolitinib or Placebo in Combination With Capecitabine in Subjects With Advanced or Metastatic Adenocarcinoma of the Pancreas Who Have Failed or Are Intolerant to First-Line Chemotherapy (The JANUS 1 Study)
Brief Title: Study of Ruxolitinib in Pancreatic Cancer Patients (Janus 1)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early based on the results of the planned interim analysis.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-362
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic pancreatic cancer; Metastatic pancreatic adenocarcinoma that is recurrent
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ruxolitinib; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ruxolitinib plus capecitabine (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: Capecitabine
- Placebo plus capecitabine (Active Comparator)
  Interventions: Drug: Placebo; Drug: Capecitabine

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablets to be administered by mouth twice daily (BID)
  Other Names: Jakafi ®; Jakavi ®
  Arms: Ruxolitinib plus capecitabine
Drug: Placebo — 5 mg tablets to be administered by mouth twice daily (BID)
  Arms: Placebo plus capecitabine
Drug: Capecitabine — 150 and 500 mg tablets to be administered by mouth twice daily (BID)

SUMMARY:
Determining the efficacy, based upon overall survival, of ruxolitinib added to capecitabine for the treatment of advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This was a randomized, double-blinded, placebo-controlled, Phase 3 study, in which approximately 310 participants with advanced or metastatic adenocarcinoma of the pancreas who have failed, or were intolerant to first-line chemotherapy, were to be randomized (1:1) to one of the following treatment groups:

* Treatment A (N = 155): Capecitabine + ruxolitinib
* Treatment B (N = 155): Capecitabine + placebo

Treatment consisted of repeating 21-day cycles. Capecitabine was self-administered for the first 14 days of each cycle, and ruxolitinib/placebo was self-administered daily for each cycle. Treatment for all participants continued as long as the regimen was tolerated, and the participant did not meet discontinuation criteria. Participants who discontinued study treatment before study termination were monitored for safety up to 30-35 days from the end of treatment. All participants were followed for survival until study termination or the safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas.
* Advanced adenocarcinoma of the pancreas that is inoperable or metastatic.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Received 1 prior chemotherapy regimen for advanced or metastatic disease (not including neoadjuvant and/or adjuvant therapy).
* ≥ 2 weeks elapsed from the completion of previous treatment regimen and participants must have recovered or be at a new stable baseline from any related toxicities.
* Radiographically measurable or evaluable disease
* Modified Glasgow Prognostic Score (mGPS) of 1 or 2 as defined below:

  1. mGPS of 1: C-reactive protein >10 mg/L and albumin ≥35 g/L
  2. mGPS of 2: C-reactive protein >10 mg/L and albumin <35 g/L

Exclusion Criteria:

* Received more than 1 prior regimen for advanced or metastatic disease.
* Ongoing radiation therapy, radiation therapy administered within 30 days of enrollment.
* Concurrent anticancer therapy (eg, chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, investigational therapy, or tumor embolization).
* Prior severe reaction to fluoropyrimidines, known dihydropyrimidine dehydrogenase deficiency (DPD), or other known hypersensitivity to active substances, including fluorouracil (5-FU), or ruxolitinib, or any of their excipients.
* Prior treatment with a JAK inhibitor for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fitzroy Dawkins, M.D., Study Director — Incyte Corporation
Locations (230):
- United States (153):
  - Avondale, Arizona
  - Chandler, Arizona
  - Gilbert, Arizona
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Surprise, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Anaheim, California
  - Bakersfield, California
  - Berkeley, California
  - Beverly Hills, California
  - Chula Vista, California
  - Covina, California
  - Downey, California
  - El Cajon, California
  - Fullerton, California
  - Gilroy, California
  - Glendale, California
  - La Mesa, California
  - Long Beach, California
  - Los Angeles, California
  - Lynwood, California
  - Modesto, California
  - Montebello, California
  - Northridge, California
  - Oceanside, California
  - Orange, California
  - Redondo Beach, California
  - San Diego, California
  - San Francisco, California
  - San Luis Obispo, California
  - Santa Ana, California
  - Santa Maria, California
  - Santa Monica, California
  - Torrance, California
  - Whittier, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Grand Junction, Colorado
  - Longmont, Colorado
  - Thornton, Colorado
  - New Britain, Connecticut
  - New Haven, Connecticut
  - Southington, Connecticut
  - Trumbull, Connecticut
  - Newark, Delaware
  - Boca Raton, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Carrollton, Georgia
  - Cartersville, Georgia
  - Douglasville, Georgia
  - Marietta, Georgia
  - Newnan, Georgia
  - Rome, Georgia
  - Thomasville, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Hinsdale, Illinois
  - Niles, Illinois
  - Urbana, Illinois
  - Goshen, Indiana
  - Indianapolis, Indiana
  - Topeka, Kansas
  - Ashland, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Scarborough, Maine
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Rockville, Maryland
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Woodbury, Minnesota
  - Bolivar, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Kalispell, Montana
  - Hastings, Nebraska
  - Omaha, Nebraska
  - Papillion, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - East Orange, New Jersey
  - Farmington, New Mexico
  - Binghamton, New York
  - Fresh Meadows, New York
  - Hudson, New York
  - Johnson City, New York
  - New York, New York
  - Nyack, New York
  - Rochester, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Wake Forest, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Columbus, Ohio
  - Middletown, Ohio
  - Oregon, Ohio
  - Toledo, Ohio
  - Eugene, Oregon
  - Portland, Oregon
  - Springfield, Oregon
  - Tualatin, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Seneca, South Carolina
  - Spartanburg, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Bedford, Texas
  - Cedar Park, Texas
  - Dallas, Texas
  - Denton, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Tyler, Texas
  - Waco, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Blacksburg, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Salem, Virginia
  - Wytheville, Virginia
  - Seattle, Washington
  - Vancouver, Washington
  - Madison, Wisconsin
- Australia (4):
  - Australian Capital Territory
  - New South Wales
  - South Australia
  - Victoria
- Belgium (8):
  - Aalst
  - Bruges
  - Brussels
  - Edegem
  - Ghent
  - Gilly
  - Kortrijk
  - Leuven
- Canada (7):
  - Calgary, Alberta
  - Oshawa, Ontario
  - Sault Ste. Marie, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Laval, Quebec
  - Montreal, Quebec
- Germany (7):
  - Aschaffenburg
  - Berlin
  - Bochum
  - Cologne
  - Essen
  - Frankford
  - Velbert
- Italy (13):
  - Aviano
  - Bari
  - Bergamo
  - Brescia
  - Cremona
  - Florence
  - Genova
  - Lido di Camaiore
  - Milan
  - Napoli
  - Pisa
  - Rimini
  - Roma
- New Zealand (3):
  - Auckland
  - Christchurch
  - Hamilton
- South Korea (3):
  - Hwasun-gun
  - Seongnam-si
  - Seoul
- Spain (5):
  - Badajoz
  - Barcelona
  - Madrid
  - Málaga
  - Seville
- Taiwan (3):
  - Taichung
  - Tainan
  - Taipei
- Thailand (3):
  - Patumwan
  - Ratchathewi
  - Seetatarom
- United Kingdom (21):
  - Aberdeen
  - Bangor
  - Birmingham
  - Boston
  - Bristol
  - Cardiff
  - Glasgow
  - Guildford
  - Harlow
  - Huddersfield
  - Lancaster
  - Leeds
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Newcastle upon Tyne
  - Nottingham
  - Plymouth
  - Southampton
  - Sutton
  - Welwyn Garden City

REFERENCES:
- [Derived] Hurwitz H, Van Cutsem E, Bendell J, Hidalgo M, Li CP, Salvo MG, Macarulla T, Sahai V, Sama A, Greeno E, Yu KH, Verslype C, Dawkins F, Walker C, Clark J, O'Reilly EM. Ruxolitinib + capecitabine in advanced/metastatic pancreatic cancer after disease progression/intolerance to first-line therapy: JANUS 1 and 2 randomized phase III studies. Invest New Drugs. 2018 Aug;36(4):683-695. doi: 10.1007/s10637-018-0580-2. Epub 2018 Mar 6. PMID 29508247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced or metastatic adenocarcinoma of the pancreas who had failed or were intolerant to first-line chemotherapy were randomized in the study.
Pre-assignment Details: Treatment was started as soon as possible after randomization (within 3 days) and consisted of continuous 21-day cycles. Capecitabine was self-administered for the first 14 days of each cycle, and ruxolitinib/placebo was self-administered for the entire cycle.
Groups:
- Ruxolitinib Plus Capecitabine: Ruxolitinib 5 mg tablets in combination with Capecitabine 150 mg or 500 mg tablets to be administered by mouth twice daily (BID).
- Placebo Plus Capecitabine: Placebo 5 mg matching placebo tablets in combination with Capecitabine: 150 mg or 500 mg tablets to be administered by mouth twice daily (BID).
Period: Overall Study
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Started | 161 | 160
Completed | 5 (Treatment ongoing as of 20APR2016 for remaining participants in the study.) | 4 (Treatment ongoing as of 20APR2016 for remaining participants in the study.)
Not Completed | 156 | 156
Not completed — Death | 13 | 8
Not completed — Adverse Event | 8 | 16
Not completed — Subject decision | 8 | 9
Not completed — Disease progression | 104 | 108
Not completed — Noncompliance with study treatment | 1 | 0
Not completed — Study terminated by the sponsor | 4 | 6
Not completed — Physician Decision | 7 | 2
Not completed — Other unspecified | 11 | 7

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine | Total
Number analyzed (Participants) | 161 | 160 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.35) | 65.6 (9.55) | 66.4 (9.48)
Age, Customized [Number; unit: participants]
  ≤ 65 years | 65 | 68 | 133
  > 65 years | 96 | 92 | 188
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 130
  Male | 95 | 96 | 191

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is reported here based on the number of deaths from randomization up to 6-months or to the data cutoff 11FEB2016.
Time Frame: Randomization until death due to any cause; up to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 161 | 160
Participants
  Observed | 113 | 124
  Censored | 48 | 36
Statistical Analysis 1: Comparison: Ruxolitinib Plus Capecitabine vs Placebo Plus Capecitabine; Test type: Other; Hazard Ratio (HR) = 0.969, 95% CI 2-sided [0.747 to 1.256]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, unequivocal progression of non-target lesions, or the appearance of new lesions.
Time Frame: Randomization to disease progression, or death due to any cause if sooner; up to 6-months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 161 | 160
days | 43.0 [41.0 to 46.0] | 44.0 [42.0 to 48.0]
Statistical Analysis 1: Comparison: Ruxolitinib Plus Capecitabine vs Placebo Plus Capecitabine; Test type: Other; Hazard Ratio (HR) = 1.056, 95% CI 2-sided [0.827 to 1.348]

3. Secondary Outcome: Percentage of Participants Achieving Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization until the earliest date of disease progression determined by investigator assessment of objective radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause if sooner. Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, unequivocal progression of non-target lesions, or the appearance of new lesions.
Time Frame: as for outcome 2
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 161 | 160
percentage of participants
  Survival rate at 3 months | 18.9 [12.7 to 25.9] | 19.8 [13.6 to 26.8]
  Survival rate at 6 months | 6.1 [2.5 to 12.2] | 5.7 [2.3 to 11.3]
  Survival rate at 9 months | 2.5 [0.5 to 7.5] | 3.4 [1.0 to 8.5]
  Survival rate at 12 months | 2.5 [0.5 to 7.5] | NA [NA to NA] — PFS was not evaluable in the placebo group due to the insufficient number of participants with events.

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate determined by radiographic disease assessments per RECIST (v1.1), by investigator assessment and was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria in Solid Tumours (RECIST) at any post baseline visit. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) : Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions with no worsening of non-target lesions and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: Baseline through end of study; up to 6-months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 161 | 160
percentage of participants
  Objective response | 3.7 | 1.9
  Complete response | 0 | 0
  Partial response | 3.7 | 1.9

5. Secondary Outcome: Duration of Response
Description: Duration of overall response was defined as the time in months from Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria in Solid Tumours (RECIST v1.1) until the first date Progressive Disease (PD) was objectively documented or until the date of death.
Time Frame: Baseline through end of study; up to 6-months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 161 | 160
days | NA [NA to NA] — The median duration of response was not evaluable in the treatment group due to the insufficient number of participants with events. | NA [NA to NA] — The median duration of response was not evaluable in the treatment group due to the insufficient number of participants with events.

6. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A treatment-emergent AE was defined as an event occurring after exposure to at least 1 dose of study drug (ruxolitinib or placebo). A treatment-related AE was defined as an event with a definite, probable, or possible causality to study medication. A serious AE is an event resulting in death, hospitalization, persistent or significant disability/incapacity, or is life threatening, a congenital anomaly/birth defect or requires medical or surgical intervention to prevent 1 of the outcomes above. The intensity of an AE was graded according to the National Cancer Institute common terminology criteria for adverse events (NCI-CTCAE) version 4.03: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (life-threatening).
Time Frame: Baseline through approximately 30 days post treatment discontinuation; up to 6-months or to the data cutoff 11FEB2016.
Population: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug (ruxolitinib or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 153 | 154
Participants
  Participants who had any TEAEs | 152 | 152
  Participants who had treatment-related TEAEs | 73 | 59
  Participants who had SAEs | 94 | 83
  Participants who had Grade 3 or higher TEAEs | 112 | 113
  Participants hospitalized because of a TEAE | 89 | 75
  Participants discontinued treatment due to TEAE | 12 | 22
  Participants with a dose modification due to TEAE | 68 | 48
  Participants on concomitant medication due to TEAE | 131 | 122
  Participants with procedure performed due to TEAE | 60 | 46
  Participants who had a fatal TEAE | 20 | 15

ADVERSE EVENTS:
Time Frame: From the first dose of study medication through study termination up to 6-months or to the data cutoff 11Feb2016.
Description: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug (ruxolitinib or placebo).
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Serious Adverse Events (participants affected / at risk) | 94/153 | 83/154
Other Adverse Events (participants affected / at risk) | 147/153 | 145/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Plus Capecitabine (N=153) | Placebo Plus Capecitabine (N=154)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 19
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 5 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Duodenal obstruction (Gastrointestinal disorders) | 2 | 3
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 5
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 7 | 4
Asthenia (General disorders) | 0 | 3
Device leakage (General disorders) | 0 | 1
Device malfunction (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 3
Hypothermia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 3 | 2
Pyrexia (General disorders) | 8 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 3
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Biloma (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 3 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2
Biliary sepsis (Infections and infestations) | 0 | 2
Biliary tract infection (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Cholangitis suppurative (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Klebsiella infection (Infections and infestations) | 2 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 7
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 5
Septic shock (Infections and infestations) | 0 | 2
Skin candida (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 4 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Failure to thrive (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 5 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 2
Phlebitis (Vascular disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Plus Capecitabine (N=153) | Placebo Plus Capecitabine (N=154)
Nausea (Gastrointestinal disorders) | 45 | 49
Anemia (Blood and lymphatic system disorders) | 45 | 22
Fatigue (General disorders) | 47 | 50
Diarrhea (Gastrointestinal disorders) | 42 | 36
Abdominal pain (Gastrointestinal disorders) | 36 | 49
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 37 | 26
Vomiting (Gastrointestinal disorders) | 30 | 46
Constipation (Gastrointestinal disorders) | 33 | 27
Stomatitis (Gastrointestinal disorders) | 30 | 18
Decreased appetite (Metabolism and nutrition disorders) | 30 | 47
Pyrexia (General disorders) | 25 | 13
Ascites (Gastrointestinal disorders) | 21 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 16
Dizziness (Nervous system disorders) | 19 | 12
Oedema peripheral (General disorders) | 18 | 35
Asthenia (General disorders) | 17 | 18
Abdominal distension (Gastrointestinal disorders) | 15 | 11
Dehydration (Metabolism and nutrition disorders) | 10 | 9
Hypotension (Vascular disorders) | 12 | 8
Abdominal pain upper (Gastrointestinal disorders) | 13 | 14
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 5
Insomnia (Psychiatric disorders) | 13 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 19
Oedema (General disorders) | 11 | 3
Urinary tract infection (Infections and infestations) | 9 | 6
Aspartate aminotransferase increased (Investigations) | 10 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Fall (Injury, poisoning and procedural complications) | 10 | 4
Weight decreased (Investigations) | 10 | 6
Alanine aminotransferase increased (Investigations) | 9 | 4
Flatulence (Gastrointestinal disorders) | 9 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Chills (General disorders) | 8 | 4
Hypertension (Vascular disorders) | 8 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 9
Dysgeusia (Nervous system disorders) | 4 | 8
Dry mouth (Gastrointestinal disorders) | 3 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 12

LIMITATIONS AND CAVEATS:
The study was terminated as other related studies of ruxolitinib did not provide sufficient efficacy to warrant continuation at the recommendation of the Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.